CLINICAL TRIAL: NCT02170415
Title: Development of a Personalised Care Plan Designed to Reduce Chronic Post-Operative Pain Following Breast Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CCR 4116
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Persistent Post-surgical Pain; Neuropathic Pain; Cancer Pain
Keywords: Persistent post-surgical pain; Breast surgery; Complex intervention; Pain treatment
MeSH Terms: conditions — Neuralgia; Cancer Pain; Agnosia | interventions — Pregabalin; Hospitals

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention limb (Active Comparator): Medical review and analgesic optimisation.
  Pain education (in the form of leaflet and website recommendations)
  Psychological input for patients with evidence of psychological morbidity.
  Protective analgesia - one pre-procedure dose of 150mg oral pregabalin.
  Five days post-procedure oral pregablin twice daily at a dose of 75mg twice a day.
  Patients offered a paravertebral block, local anaesthetic infiltrated around the wound by the surgeon.
  Daily, focused visits from the hospital pain team.
  Any patient displaying concerning pain symptoms, behaviour or who underwent prolonged (>3 hours surgery) may be booked for early 'preemptive' review in pain clinic.
  Interventions: Drug: Protective analgesia; Other: Pain education; Behavioral: Psychological support; Procedure: Paravertebral block/local anaesthetic infiltration; Other: Daily visits from pain team whilst in hospital
- Usual care (No Intervention): These partcipants will receive usual care before, during and after their breast surgery

INTERVENTIONS:
Drug: Protective analgesia — Participants in the intervention arm of the study (if no contraindications exist) will be administered one pre-procedure dose of 150mg of oral pregabalin.
  For a total of five days post-procedure the participants in the intervention limb of the study will take oral pregablin twice daily at a dose of 75mg twice a day.
  Other Names: Pregabalin
  Arms: Intervention limb
Other: Pain education — Participant will receive a pain education leaflet
  Arms: Intervention limb
Behavioral: Psychological support — Participants demonstrating psychological morbidity will be offered psychological support prior to surgery
  Arms: Intervention limb
Procedure: Paravertebral block/local anaesthetic infiltration — Patients on the intervention limb will be encouraged to have a paravertebral block if not contraindicated
  Arms: Intervention limb
Other: Daily visits from pain team whilst in hospital
  Arms: Intervention limb

SUMMARY:
Numerous surveys have shown that following breast surgery, longterm pain affects around half of patients. Given that 1 in 9 women will get breast cancer and that surgery is the cornerstone of treatment, persistent pain represents a major challenge. In addition to the suffering chronic pain causes to individual patients, the investigators know that it places a substantial burden on families and carers, and that patients with pain represent an excessive demand on healthcare resources.

This research will evaluate the impact of introducing a proactive, integrated care plan for patients having breast surgery. It will assess the effect of the care plan on reducing the number of patients with pain at 3 and 12 months after their procedure.

The personalised plan involves numerous evidence based steps linked by a single unifying description aimed at controlling pain, before, during and after the procedure, in hospital and at home.

Patients at risk of developing pain will be identified prior to the procedure and randomly allocated to follow either the personalised care plan or to receive 'usual' care. In the personalised care plan group, participants will get information about chronic pain, be screened for pain and offered immediate treatment. During their procedure both the surgeon and the anaesthetist will offer treatments such as nerve numbing procedures that reduce the likelihood of experiencing pain.

After their procedure, patients will be again screened for pain and further treatment instigated. Physiotherapists and other allied health professionals such as psychologists will also be involved as appropriate. A package of care for pain will then be passed on to the patients' GP, in the form of a written pain management plan, for ongoing care which will be linked to the hospital. Patients from both groups will be followed up for a year at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 and over with breast cancer undergoing breast surgery at the Royal Marsden Hospital. This includes mastectomy, wide local excision with axillary clearance, breast reconstruction surgery i.e Diep flap, LD flap

Exclusion Criteria:

* Previous thoracic surgery.
* Symptomatic angina pectoris.
* Renal impairment.
* Inability to read or to understand consent documentation.
* Patients undergoing the following surgery; lumpectomy, wide local excision, cosmetic procedures, any day-case breast surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Difference in pain scores (as indicated by a pain severity index score) in the intervention group compared to the 'usual care' group. | 3 months

SECONDARY OUTCOMES:
The difference in levels of anxiety and depression (versus 'usual care') measured by the hospital anxiety and depression scale (HADS) | 3 and 12 months
The difference in general health outcomes (versus 'usual care') determined by the EQ5D questionnaire | 3 and 12 months
The difference in participant satisfaction (versus 'usual care') determined by the Global Surgical Recovery (GSR) Scale. | 3 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: JOHN E WILLIAMS, MB BS FRCA, Principal Investigator — The Royal Marsden Hospital
Locations (1):
- The Royal Marsden Hospital, London, London, United Kingdom